CLINICAL TRIAL: NCT03758820
Title: Multicenter Study, Randomized, Parallel Group Controlled, Testing the Effectiveness of a Behavioral Cognitive Therapy (BCT) vs Usual Local Practice on the Fatigue of Patients With Relapsing Remittent Multiple Sclerosis (RRMS)
Brief Title: Behavior Cognitive Therapy on Fatigue Impact in MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Réseau Sep Idf Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FACCSEP
Record Dates: First submitted 2017-10-19; First posted 2018-11-29 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Fatigue; Cognitive Therapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue

STUDY DESIGN:
Intervention Model Description: parallel group assignment
Who Masked: Participant
Masking Description: randomization of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCT group (Experimental): Intervention : Behavorial Cognitive Therapy (BCT) will be delivered by two psychologists at six once-weekly sessions of 90 minutes (with homework activities between the sessions) + 4 booster sessions at week 6, 12, 18 and 36 after the end of the programme.
  It was designed for groups of 8 to 10 people. The programme is standardised: PowerPoints presentations support each session and a detailed facilitator manual and companion patient workbook. accompany the programme.
  Interventions: Behavioral: Behavorial Cognitive Therapy (BCT)
- Control group (No Intervention): Usual local practice

INTERVENTIONS:
Behavioral: Behavorial Cognitive Therapy (BCT) — Check-in : review of the homewok Talk : Presentation of the aim of the session Group Activity : Relaxation and Execises Refreshment break Homework : exercises to practice at home and explanation about the forms to fill in.
  Passout : session handbook and supports for exercises.
  Arms: BCT group

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease that leads to demyelination of the central nervous system. Fatigue is one of the most frequent and most disabling symptoms of MS. Up to 86% of individuals with MS experience fatigue at any one time; 65% consider it to be one of their three most troubling symptoms. Fatigue may limit or prevent participation in dayly activities and reduce psychological well-being (1, 2). Pharmacological and non-pharmacological treatments are available for MS-related fatigue, but evidence on effectiveness is mostly inconclusive or non-existent. The psychological approaches of fatigue management are interesting. To date, three RCTs using cognitive-behavioral group-based approaches in MS fatigue management programs have demonstrated their effectiveness (3-6). The results demonstrated a reduction in fatigue scores and better self-management of the disease in general. However, if these programs are effective at the time of their application and in the medium term, the issue of maintaining long-term therapeutic benefits is problematic.

The aim of this research is to assess the effectiveness of the FACETS program (6), on a population of French patients with RRMS over a 18 month period. This program focuses on the management of fatigue and is based on a conceptual framework that incorporates elements of cognitive-behavioral, self-efficacy, self-management and energy effectiveness theories. It consists of six once-weekly sessions of 90 minutes, with homework activities between the sessions. It is designed for groups of 6 to 10 people. The investigators propose to add 4 booster sessions to the FACETS program, at week 6, 12, 18 et 36 after the end of the program, in order to activate and reinforce the cognitive and behavioral processes and enhance the benefits of FACETS in the longer term.

This trial is randomized controlled comparative comparing a group receiving a FACETS program with a group receiving only a current local practice. Socio-demographic and medical data are measured as well as fatigue impact, fatigue severity, anxiety and depression, sleep disorder and quality of life.

The expected results are a significantly greater decrease in fatigue severity and impact in the FACETS group than the control group post intervention and this difference will be maintained at 1 year.

DETAILED DESCRIPTION:
In spite of the fatigue impact is well known in MS, medical care of this symptom is not usual. Moreover, treatments of fatigue are available, but evidence for effectiveness is limited. This study will build upon the existing evidence base for the effectiveness of cognitive behavioral approaches, and particularly the recent FACETS trial published by co-applicants.

Scientific aim is to assess the effectiveness of the FACETS program plus 4 additional booster sessions on a population of French patients with RRMS over a 12 months period.

This study will provide evidence on whether the FACETS program plus booster sessions is effective in helping MS patients with their fatigue. The program is designed to facilitate use within health services. Thus, if the results from this trial are positive, there is potential for directly adding to the treatment options available to MS patients who have troublesome fatigue, and improving the central nervous system affecting approximately 2.5 million people (5). Fatigue is one of the most commonly reported and disabling symptoms of MS, often occurring daily (6) and with a variable course (7-8). Up to 86% of individuals with MS experience fatigue at any one time; 65% consider it to be one of their three most troubling symptoms. Fatigue has been defined as a "subjective lack of physical and/or mental energy that is perceived by the individual or caregiver to interfere with usual or desired activities" (9).

Researchers have distinguished between primary and secondary fatigue (10). "Primary" fatigue relates to aspects of fatigue deemed to be directly related to the disease process such as lassitude or asthenia (an overwhelming sense of tiredness not directly related to participation in activity or exercise), "short-circuiting" fatigue (when muscular performance deteriorates during sustained activity but recovers after a short rest break) and heat sensitive fatigue (where fatigue is triggered or worsened by heat). "Secondary" fatigue refers to fatigue that is not unique to MS and is related to factors common to a range of chronic and disabling conditions (e.g. sleep disturbance, medication side effects, infection, physical exertion, depression, anxiety, stressful life events, characteristics of the local environment - such as lighting and temperature within a work setting). The relationship between these dimensions is complex; various symptoms of MS may act as predisposing factors for secondary fatigue.

Fatigue may limit or prevent participation in everyday activities, work, leisure and social pursuits, restrict role fulfilment and reduce psychological well-being (1-2) and is one of the key precipitants of early retirement (11-12). Its 'invisible' nature may lead to difficulties in personal and work relationships (13-14).

Although fatigue is one of the major symptoms of MS patients, the pathophysiology of fatigue is unclear (15) but likely to be multi- factorial (16-17). Findings on the relationships between fatigue and other clinical variables (such as age, gender, disease duration, and clinical activity) have been equivocal (18). The neural correlates are poorly components such as peripheral vs. central fatigue or physical vs. cognitive or mental, which are difficult to define or operationalize.

Pharmacological and non-pharmacological treatments are available for MS-related fatigue, but evidence on effectiveness is mostly inconclusive or non-existent (19-20). Non-pharmacological studies exploring the effectiveness of energy conservation programs for MS-fatigue have tended to be small and uncontrolled (21-22). Although the important relationships between physical and psychological aspects of MS-fatigue are recognized, high quality randomized and controlled trials (RCTs) of psychological interventions are rare (23).

The integration of cognitive-behavioral approaches in fatigue management programs is interesting. Indeed, their effectiveness has been demonstrated in Chronic Fatigue Syndrome. To date, three RCTs using cognitive-behavioral group-based approaches in the context of MS have been conducted (3-4). Cognitive behavioral approaches are potentially more profitable than the dual interventions, more easily integrated into a framework of routine care, and they also offer the possibility of peer support. The results of these studies demonstrated a reduction in fatigue scores and better self-management of the disease in general, resulting in improvements in quality of life. In their meta-analysis (24) indicate that the results obtained with CBT or with physical exercises are similar, but when people are anxious or depressed, which is often the case with MS (25-26), CBT shows better improvement. Knoop & al. (27) highlighted the importance of cognitive representations on fatigue and the potential relevance of CBT: they showed that the strongest mediators of fatigue severity were fatigue avoidance, symptom focusing and the belief that fatigue symptoms are a sign of damage.

Thomas et al., (4) found that modest effects on fatigue severity were largely maintained at one year (unpublished data). Given that MS typically is diagnosed during the most productive years of individuals' lives and lasts the life course it is important to give people flexible tools and strategies to manage fatigue that can be used in the long term. Booster session might therefore help to 'boost' or enhance the effectiveness of the program in the longer term Methodology A multicentre parallel arm randomized controlled trial comparing a group receiving 'enhanced' FACETS plus current usual practice versus a group receiving current local practice only.

Inclusion criteria: clinically confirmed diagnosis of relapsing remitting MS; Significant fatigue levels (score at the Modified Fatigue Impact Scale - MFIS > 45); Expanded Disability Status Scale score < 6; age ≥ 18 years; written informed consent; speak and understand French; be able to follow the program.

Exclusion criteria: Individuals with cognitive deficits such that they would not be able to engage and benefit from this group-based program. Indeed, if individuals have significant cognitive deficits, most of the content of the fatigue management program would not be appropriate; People who have had a relapse within the past three months: (a relapse might result in increased fatigue) People who have started treatment on a disease modifying drug or anti-depressant in the past 3 months (one of the possible initial side effects of these drugs is fatigue); People who have psychiatric disorders Sample size: if one uses the results of the study (30) (matched groups), these authors show that in 59 MS patients treated with Modafinil, the mean fatigue score on the MFIS is 52.3 (SD/SE = 18.5), whilst in 56 MS patients treated by placebo the mean fatigue score is 49.2 (SD/SE = 16.6). The investigators will seek to uncover an absolute difference of 10 points between mean scores. The FACETS trial found a standardized effect size of 0.35 on their fatigue severity primary outcome, which would translate to around 6 points on the MFIS. It is anticipated that by using booster sessions and by running the programme using psychologists, that the anticipated effect size will be larger (10 points). In order to detect a 10 points absolute difference between the mean scores (on the MFIS) of the efficaciousness of the cognitive-behavioral intervention, power to detect an effect size of 8.5 points Participants will be identified and recruited by the neurologists of the hospitals who take part in the program, when they come for a medical examination.

Randomization: After giving their informed consent, the patients will be entered onto the trial database and randomized in a 1:1 ratio to either the fatigue management program and or current local practice using a computer, generated randomization sequence stratified by site.

Intervention FACETS (4). Focuses on the management of fatigue and is based on a conceptual framework that incorporates elements of cognitive-behavioral, self-efficacy, self-management and energy effectiveness theories. It consists of six once-weekly sessions of 90 minutes (with a break), with homework activities between the sessions. It is designed for groups of 8 to 10 people and will be delivered by two psychologists. The program is standardized: PowerPoints presentations support each session and a detailed facilitator manual and companion patient workbook. accompany the program.

The investigators propose to add 4 booster sessions to the FACETS program, at week 6, 12 et 18 et 36 after the end of the program, in order to activate and reinforce the cognitive and behavioral processes and they hope to enhance the benefits of FACETS in the longer term.

Measures For the FACETs group these will be administered pre, post and 12 months after the end of the FACETS program and at the same times for those in the control group Socio-demographic and medical data: age, sex, level of education, marital status, number of children and professional status; date of diagnosis, disease type, level of disability.

Neuropsychological measures: Paced Auditory Serial Addition Task (PASAT,28) & the Computerized Speed Cognitive Test (CSCT,29).

Statistical analysis: They will register the trial and endeavor to publish the full trial protocol prior to its commencement. The primary analysis of effectiveness will use an "intention-to-treat" approach and focus on comparing MFIS at 12 months post treatment (ie after the program and all booster sessions are complete) between the two trial arms using analysis of covariance to take into account MFIS at baseline, and study center. In addition to these analyses they will conduct further comparative analyses using a mixed model approach that permits analysis of repeated measures (baseline, post treatment and 12 months follow-up), takes into account missing data (i.e. model allows participants to contribute to the model even if they don't have complete data), and takes into account the group-based nature of the program (cluster effects). A similar approach will be used for other interval scaled outcome measures, and adapted if the outcome measure is nominal (eg the EDSS) Hypotheses There will be a significantly greater decrease in fatigue severity and impact in the FACETS group than the control group post intervention and this difference will be maintained at 1 year.

There will be a significantly greater improvement in sleepiness and sleep quality, anxiety, depression, stress, attention and working memory in the FACETS group than the control group at the end of the program and at 12 months The FACETS group will show a significantly greater reduction in cortical atrophy, axonal loss and demyelination within white matter tracts of DMN than those in the control group Ethics The protocol was submitted to the French competent authorities and a declaration was made to the CNIL.

Patients allocated to the control group (current local practice) will be offered the FACETS program after the 12 months follow-up.

Finally, all information collected will be strictly confidential. Identification numbers of participants will be noted on the questionnaires which will not contain any names or details to identify the participants. Only members of the research team will be allowed to access the trial data.

ELIGIBILITY:
Inclusion Criteria:

* RRMS
* EDSS ≤ 5,5
* MFIS score > 45
* Outpatient treatment
* Enable to follow the BCT sessions
* French understanding
* More than 18 years old
* Inform consent signature
* Membership in a social protection

Exclusion criteria

* Cognitive disorders avoiding patient participation
* Relapse within last 3 months before baseline
* Onset of DMT within 3 months
* Onset of antidepressive treatment within 3 months
* Onset of treatment for fatigue within 3 months
* Psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change assessment from Baseline measure of Fatigue Impact to month 6, 12 and 18 | After 6 weeks and 6,12 and 18 months
  Fatigue impact evaluated by MFIS autoquestionnaire MFIS : Modified Fatigue Impact Scale, 5 response option (0 to 4), score of between 0 (better) and 84 (worse) : A score > 45 means the patient is affected by fatigue.

SECONDARY OUTCOMES:
Change assessment from Baseline of Anxiety and depression | After 12 months
  Anxiety and depression evaluated by HADS autoquestionnaire HADS : Hospital Anxiety and Depression Scale, five-point rating scale (0 to 4), score of between 0 (better) and 42 (worse).
Change assessment from Baseline of Fatigue severity | After 6 weeks and 6 and 12 months
  Fatigue severity evaluated by FSS autoquestionnaire FSS : Fatigue Severity Scale, seven-point rating scale (1 to 7), score >3 = fatigue severity
Change assessment from Baseline of Quality of sleep: Pittsburgh Sleep Quality scale | After 12 months
  Quality of sleep evaluated by Pittsburgh scale. IQSP 1.0 : Pittsburgh Sleep Quality scale, four-point rating scale (0 to 3), score of between 0 (better) and 21 (worse) : score >5 = sleep disorder.
Change assessment from Baseline of Quality of sleep: Epworth Sleepiness Scale | After 12 months
  Quality of sleep evaluated by Epsworth scale. Epworth Sleepiness Scale : four-point rating scale (0 to 3), score of between 0 (better) and 24 (worse) : score >9 = risk of pathological somnolence
Change assessment from Baseline of Cognitive disorders | After 12 months
  Cognitive disorders evaluated by PASAT. PASAT : Paced Auditory Serial Addition Test de Gronwall. Score of between 0 (worse) and 60 (better).
Change assessment from Baseline of Cognitive disorders | After 12 months
  Cognitive disorders evaluated by CSCT. CSCT : Computerized speed cognitive test. The score is the number of correct answer provided in 90 seconds. At the end of each test, the patient's score is automatically interpreted according to the normative values for his age, level of education and sex. If a patient's score is less than 1.5 SD of normal values, it is likely that this patient has a TTI slowing.
Change assessment from Baseline of Quality of life: MSIS-29 | After 6,12 and 18 months
  Quality of life evaluated by MSIS-29. MSIS-29 : The Multiple Sclerosis Impact Scale. 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. 5 response options (1 to 5). Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
Change assessment from Baseline of Quality of life: EQ5D-3L | After 6,12 and 18 months
  Quality of life evaluated by EQ5D-3L. EQ5D-3L European Quality of Life. Five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change assessment from Baseline of Medical care consumption and professional impact | After 6,12 and 18 months
  Medical care consumption evaluated by the number of visits to the physician, treatment and hospitalization
Change assessment from Baseline of professional impact | After 6,12 and 18 months
  professional impact evaluated by the number of work stoppage

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HEINZLEF, MD, Principal Investigator — Réseau Sep Idf Ouest
Locations (1):
- Poissy St Germain Hospital, Poissy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edgley KJ. Sullivan M, Dehoux E. A survey of multiple sclerosis: II. Determinants of employment status. Can J Rehabil 4:127-132, 1991
- [Background] Multiple Sclerosis Council. Fatigue and Multiple Sclerosis - Clinical Practice Guidelines, 1998.
- [Background] Bowcher H, May M. Occupational Therapy for the Management of Fatigue in Multiple Sclerosis, Br J Occup Ther, 61(11):488-492, 1998.
- [Background] Castell BD, Kazantzis N, Moss-Morris RE. Cognitive Behavioral Therapy and Graded Exercise for Chronic Fatigue Syndrome: A Meta-Analysis. Clin Psychol Sci Pract. 18(4):311-324, 2012.
- [Result] Amato MP, Ponziani G, Siracusa G, Sorbi S. Cognitive dysfunction in early-onset multiple sclerosis: a reappraisal after 10 years. Arch Neurol. 2001 Oct;58(10):1602-6. doi: 10.1001/archneur.58.10.1602. PMID 11594918
- [Result] van Kessel K, Moss-Morris R, Willoughby E, Chalder T, Johnson MH, Robinson E. A randomized controlled trial of cognitive behavior therapy for multiple sclerosis fatigue. Psychosom Med. 2008 Feb;70(2):205-13. doi: 10.1097/PSY.0b013e3181643065. Epub 2008 Feb 6. PMID 18256342
- [Result] Thomas S, Thomas PW, Kersten P, Jones R, Green C, Nock A, Slingsby V, Smith AD, Baker R, Galvin KT, Hillier C. A pragmatic parallel arm multi-centre randomised controlled trial to assess the effectiveness and cost-effectiveness of a group-based fatigue management programme (FACETS) for people with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1092-9. doi: 10.1136/jnnp-2012-303816. Epub 2013 May 21. PMID 23695501
- [Result] Compston A, Coles A. Multiple sclerosis. Lancet. 2002 Apr 6;359(9313):1221-31. doi: 10.1016/S0140-6736(02)08220-X. PMID 11955556
- [Result] Branas P, Jordan R, Fry-Smith A, Burls A, Hyde C. Treatments for fatigue in multiple sclerosis: a rapid and systematic review. Health Technol Assess. 2000;4(27):1-61. PMID 11074395
- [Result] Johansson S, Ytterberg C, Hillert J, Widen Holmqvist L, von Koch L. A longitudinal study of variations in and predictors of fatigue in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):454-7. doi: 10.1136/jnnp.2007.121129. PMID 18344396
- [Result] Debouverie M, Pittion-Vouyovitch S, Guillemin F. [Reconsidering fatigue at the onset of multiple sclerosis]. Rev Neurol (Paris). 2009 Mar;165 Suppl 4:S135-44. doi: 10.1016/S0035-3787(09)72125-3. French. PMID 19361678
- [Result] Monks J. Experiencing symptoms in chronic illness: fatigue in multiple sclerosis. Int Disabil Stud. 1989 Apr-Jun;11(2):78-83. doi: 10.3109/03790798909166394. PMID 2630556
- [Result] Grima DT, Torrance GW, Francis G, Rice G, Rosner AJ, Lafortune L. Cost and health related quality of life consequences of multiple sclerosis. Mult Scler. 2000 Apr;6(2):91-8. doi: 10.1177/135245850000600207. PMID 10773854
- [Result] Flensner G, Landtblom AM, Soderhamn O, Ek AC. Work capacity and health-related quality of life among individuals with multiple sclerosis reduced by fatigue: a cross-sectional study. BMC Public Health. 2013 Mar 15;13:224. doi: 10.1186/1471-2458-13-224. PMID 23497281
- [Result] White LJ, Castellano V. Exercise and brain health--implications for multiple sclerosis: Part 1--neuronal growth factors. Sports Med. 2008;38(2):91-100. doi: 10.2165/00007256-200838020-00001. PMID 18201113
- [Result] Ritvo PG, Fisk JD, Archibald CJ, Murray TJ, Field C. Psychosocial and neurological predictors of mental health in multiple sclerosis patients. J Clin Epidemiol. 1996 Apr;49(4):467-72. doi: 10.1016/0895-4356(95)00027-5. No abstract available. PMID 8621999
- [Result] Schwid SR, Covington M, Segal BM, Goodman AD. Fatigue in multiple sclerosis: current understanding and future directions. J Rehabil Res Dev. 2002 Mar-Apr;39(2):211-24. PMID 12051465
- [Result] Racke MK, Hawker K, Frohman EM. Fatigue in multiple sclerosis: is the picture getting simpler or more complex? Arch Neurol. 2004 Feb;61(2):176-7. doi: 10.1001/archneur.61.2.176. No abstract available. PMID 14967763
- [Result] Bakshi R. Fatigue associated with multiple sclerosis: diagnosis, impact and management. Mult Scler. 2003 Jun;9(3):219-27. doi: 10.1191/1352458503ms904oa. PMID 12814166
- [Result] Kos D, Kerckhofs E, Nagels G, D'hooghe MB, Ilsbroukx S. Origin of fatigue in multiple sclerosis: review of the literature. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):91-100. doi: 10.1177/1545968306298934. Epub 2007 Apr 4. PMID 17409388
- [Result] Tejani AM, Wasdell M, Spiwak R, Rowell G, Nathwani S. Carnitine for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD007280. doi: 10.1002/14651858.CD007280.pub2. PMID 20166093
- [Result] Vanage SM, Gilbertson KK, Mathiowetz V. Effects of an energy conservation course on fatigue impact for persons with progressive multiple sclerosis. Am J Occup Ther. 2003 May-Jun;57(3):315-23. doi: 10.5014/ajot.57.3.315. PMID 12785670
- [Result] Mathiowetz VG, Finlayson ML, Matuska KM, Chen HY, Luo P. Randomized controlled trial of an energy conservation course for persons with multiple sclerosis. Mult Scler. 2005 Oct;11(5):592-601. doi: 10.1191/1352458505ms1198oa. PMID 16193899
- [Result] Lee MA, Smith S, Palace J, Matthews PM. Defining multiple sclerosis disease activity using MRI T2-weighted difference imaging. Brain. 1998 Nov;121 ( Pt 11):2095-102. doi: 10.1093/brain/121.11.2095. PMID 9827769
- [Result] Gay MC, Vrignaud P, Garitte C, Meunier C. Predictors of depression in multiple sclerosis patients. Acta Neurol Scand. 2010 Mar;121(3):161-70. doi: 10.1111/j.1600-0404.2009.01232.x. Epub 2010 Jan 12. PMID 20070277
- [Result] Feinstein A, Magalhaes S, Richard JF, Audet B, Moore C. The link between multiple sclerosis and depression. Nat Rev Neurol. 2014 Sep;10(9):507-17. doi: 10.1038/nrneurol.2014.139. Epub 2014 Aug 12. PMID 25112509
- [Result] Knoop H, van Kessel K, Moss-Morris R. Which cognitions and behaviours mediate the positive effect of cognitive behavioural therapy on fatigue in patients with multiple sclerosis? Psychol Med. 2012 Jan;42(1):205-13. doi: 10.1017/S0033291711000924. Epub 2011 Jun 15. PMID 21672300
- [Result] Gronwall DM. Paced auditory serial-addition task: a measure of recovery from concussion. Percept Mot Skills. 1977 Apr;44(2):367-73. doi: 10.2466/pms.1977.44.2.367. PMID 866038
- [Result] Ruet A, Deloire MS, Charre-Morin J, Hamel D, Brochet B. A new computerised cognitive test for the detection of information processing speed impairment in multiple sclerosis. Mult Scler. 2013 Oct;19(12):1665-72. doi: 10.1177/1352458513480251. Epub 2013 Mar 4. PMID 23459569
- [Result] Stankoff B, Waubant E, Confavreux C, Edan G, Debouverie M, Rumbach L, Moreau T, Pelletier J, Lubetzki C, Clanet M; French Modafinil Study Group. Modafinil for fatigue in MS: a randomized placebo-controlled double-blind study. Neurology. 2005 Apr 12;64(7):1139-43. doi: 10.1212/01.WNL.0000158272.27070.6A. PMID 15824337
- [Derived] Gay MC, Cassedanne F, Barbot F, Vaugier I, Thomas S, Manchon E, Bensmail D, Blanchere M, Heinzlef O. Long-term effectiveness of a cognitive behavioural therapy (CBT) in the management of fatigue in patients with relapsing remitting multiple sclerosis (RRMS): a multicentre, randomised, open-label, controlled trial versus standard care. J Neurol Neurosurg Psychiatry. 2024 Jan 11;95(2):158-166. doi: 10.1136/jnnp-2023-331537. PMID 37648439